CLINICAL TRIAL: NCT02802917
Title: Evaluation of the Stinging Potential of Products in Human Eyes
Brief Title: To Evaluate Eye Installation-Tear Free
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18271
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agents
Keywords: Eye stinging potential

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SPF 50 Y49 091 (Experimental): Subjects were given the control article (standard shampoo mixture, X46 046) in one eye and one of the test articles in the other eye according to the randomization schedule.
  Interventions: Drug: SPF 50 Y49 091 (BAY 987516); Other: J & J baby shampoo, X46 046 (control)
- SPF 50 X15 158 (Experimental): Subjects were given the control article (standard shampoo mixture, X46 046) in one eye and one of the test articles in the other eye according to the randomization schedule.
  Interventions: Drug: SPF 50 X15 158 (BAY 987516); Other: J & J baby shampoo, X46 046 (control)
- SPF 50 X15 160 (Experimental): Subjects were given the control article (standard shampoo mixture, X46 046) in one eye and one of the test articles in the other eye according to the randomization schedule.
  Interventions: Drug: SPF 50 X15 160 (BAY 987516); Other: J & J baby shampoo, X46 046 (control)
- SPF 50 X57 162 (Experimental): Subjects were given the control article (standard shampoo mixture, X46 046) in one eye and one of the test articles in the other eye according to the randomization schedule.
  Interventions: Drug: SPF 50 X57 162 (BAY 987516); Other: J & J baby shampoo, X46 046 (control)

INTERVENTIONS:
Drug: SPF 50 Y49 091 (BAY 987516) — 5 μL of the appropriate test or control article were instilled into the lower conjunctival sac of the eye.
  Arms: SPF 50 Y49 091
Drug: SPF 50 X15 158 (BAY 987516) — 5 μL of the appropriate test or control article were instilled into the lower conjunctival sac of the eye.
  Arms: SPF 50 X15 158
Drug: SPF 50 X15 160 (BAY 987516) — 5 μL of the appropriate test or control article were instilled into the lower conjunctival sac of the eye.
  Arms: SPF 50 X15 160
Drug: SPF 50 X57 162 (BAY 987516) — 5 μL of the appropriate test or control article were instilled into the lower conjunctival sac of the eye.
  Arms: SPF 50 X57 162
Other: J & J baby shampoo, X46 046 (control) — 5 μL of the appropriate test or control article were instilled into the lower conjunctival sac of the eye.

SUMMARY:
The primary objective of this study was to compare the human eye stinging potential of experimental formulas of sun care products [Sun Protection Factor (SPF) 50 Y49 091, SPF 50 X15 158, SPF 50 X15 160 and SPF 50 X57 162 compared to an industry standard shampoo mixture.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, 18 to 60 years with no medical conditions of the eyes as determined by the subject's medical history and confirmed by an ophthalmologist
* Subjects not under any doctor's care for ocular or peri orbital diseases
* The subject will refrain from using contact lenses, any topical facial products, any eye drops, false eyelashes, make up, over the counter products, or cosmetics on their eyes, eyelids, eyelashes, or the periorbital areas of the face during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2015-05-24 (Actual); Study Completion 2015-05-24 (Actual)

PRIMARY OUTCOMES:
Subjective discomfort | up to 10 days
  Score 0: No discomfort felt Score 1: Faint, barely perceptible discomfort Score 2: Mild, low intensity discomfort that does not prevent the subject from opening lids Score 3: Moderately intense discomfort that interferes with but does not prevent lid opening Score 4: Severe, very intense discomfort that makes voluntary lid opening difficult, requires force to pull lids apart, and results in the subject requesting washout of test article
Objective lacrimation | up to 10 days
  Score 0: No tearing or lid wetness above normal Score 1: Noticeable increase in moistness of lid edges - no frank tearing Score 2: Frank tearing - meager flow Score 3: Frank tearing - moderate flow Score 4: Frank tearing - copious flow
Objective conjunctival inflammation | up to 10 days
  Score 0: Inflammatory changes absent Score 1: Capillaries slightly more prominent than they were at time of baseline examination Score 2: Capillaries very prominent plus some diffuse conjunctival reddening Score 3: Vessels very prominent plus diffuse and confluent intense redness Score 4: Beefy redness and everted lids
Objective cornea and iris inflammation | up to 10 days
  Score 0: No effect detected with use of slit lamp Score 1: Barely perceptible clouding or pitting of cornea or thickening of iris detected via slit lamp Score 2: Faint clouding or pitting of cornea and/or thickening of the iris Score 3: Moderate clouding or pitting of cornea and/or thickening of the iris Score 4: Intense clouding or pitting of cornea and/or thickening of the iris

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States